CLINICAL TRIAL: NCT03946306
Title: Comparative Evaluation of Postoperative Pain,Periapical Damage and Bacterial Disinfection After Using Endodontic Needle and Eddy Tips During Root Canal Irrigation
Brief Title: Evaluation of Postoperative Pain With Eddy Tips (EPPET)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EDDYSP; 2019-001705-24 (EudraCT Number)
Record Dates: First submitted 2019-04-23; First posted 2019-05-10 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2020-10

CONDITIONS: Pain, Postoperative
Keywords: ENDODONTIC IRRIGATION, ENDODONTIC DISINFECTION, EDDY TIPS, APICAL EXTRUSION, ENDODONTIC PAIN
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: The patients will be divided in 2 groups: Group 1: (control group) 5,25% NaOCl with syringe needle irrigation alone. Group 2: 5,25% NaOCl with syringe needle irrigation, activated with sonic system EDDY (VDW, Munich, Germany)
Who Masked: Participant
Masking Description: The patients will not know which treatment they will receive
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): 5,25% NaOCl with syringe needle irrigation alone
  Interventions: Drug: 5,25% NaOCl with syringe needle irrigation alone
- Group 2 (Active Comparator): 5,25% NaOCl with syringe needle irrigation, activated with sonic system EDDY (VDW, Munich, Germany)
  Interventions: Device: EDDY

INTERVENTIONS:
Drug: 5,25% NaOCl with syringe needle irrigation alone — In group 1 (control group), a final irrigation will be made with 1.5 ml of NaOCl per canal, during 30 seconds in an up-and-down motion, with the needle 1 mm short of the working length, without binding. After this, a 30 seconds pause will be done. This step will be repeated once again.
  Other Names: NaOCl
  Arms: Group 1
Device: EDDY — In group 2, a final irrigation will be made with 1.5 ml of NaOCl per canal and the irrigant will be activated using EDDY tips, 1 mm short of the working length without binding. The activation will be performed during 30 seconds, followed by a 30 seconds pause, and the cycle will be repeated once again, according to manufacture instructions.
  Other Names: EDDY + NaOCl
  Arms: Group 2

SUMMARY:
This investigation will focus on the use of EDDY tips, because it is known that the complete debridement of the canal is very difficult, which leads to an accumulation of tissue debris, bacteria and their products, resulting in persistent periradicular inflammation. So, it's of great importance, the study of other approaches of cleaning and disinfecting the root canal, which at the same time, may produce a lower risk of postoperative pain.

The above mentioned topics have never been analysed simultaneously with the use of EDDY tips, and the evaluation of the postoperative pain was never addressed.

This research is of great clinical interest, due to the complexity of root canal system, with isthmuses, ramifications and dentinal tubules, that make the total elimination of bacteria impossible, even with the best clinical protocols, because the irrigants cannot penetrate the dentinal tubules, and the postoperative pain is an exhausting factor for patients.

Therefore, a new protocol, with better disinfection rate and less postoperative pain, will be able to increase the success rate of endodontic treatments, allowing to save condemned teeth.

DETAILED DESCRIPTION:
CLINICAL STUDY:

1. Rate of postoperative pain of 2 endodontic disinfection protocols.

-A clinical study will be carried out, in patients that attend the Faculdade de Medicina Dentária Dental Clinic at Universidade do Porto, for initial nonsurgical root canal treatments. About 80 single-rooted and premolar teeth with mature, fully formed apices and diagnosed with irreversible pulpitis will be selected.

Patients will be excluded if they were <12 years of age; pregnant; had an indication for antibiotic prophylaxis; uncontrolled hypertension or diabetes mellitus; chronic renal failure; hematologic diseases; HIV; osteoporosis treated with bisphosphonates; steroid therapy >5mg/day of prednisolone and prior to head and neck irradiation therapy. We will also exclude teeth with abnormal root canal anatomy, with more than 26mm in length and with advanced periodontal disease. Those patients will be divided in 2 groups: Group 1: (control group) 5,25% NaOCl with syringe needle irrigation alone. Group 2: 5,25% NaOCl with syringe needle irrigation, activated with sonic system EDDY (VDW, Munich, Germany)

All the patients will receive anaesthetic solution and after anaesthesia, each tooth will be isolated using rubber dam and the access cavity will be made.

The glide path will be determined using stainless steel hand files, confirmed by periapical radiographs. The root canals will be instrumented, confirming the apical patency with a size 15 K-file, and then the instrumentation sequence. The apical patency will be maintained throughout the shaping procedure using #10 k-file between each instrument.

* All the canals will be irrigated continuously with 5,25% NaOCl during the instrumentation, with a conventional endodontic syringe with 27 gauge needle. In group 1 (control group), a final irrigation will be made with 1.5 ml of NaOCl per canal, during 30 seconds in an up-and-down motion, with the needle 1 mm short of the working length, without binding. After this, a 30 seconds pause will be done. This step will be repeated once again. In group 2, a final irrigation will be made with 1.5 ml of NaOCl per canal and the irrigant will be activated using EDDY tips, 1 mm short of the working length without binding. The activation will be performed during 30 seconds, followed by a 30 seconds pause, and the cycle will be repeated once again, according to manufacture instructions.
* After the final irrigation protocol, all the canals will be dried and sterile cotton pellets will be placed in the pulp chamber with a provisional restoration. No intracanal medicament will be placed. The obturation will be executed in the following appointment.

ELIGIBILITY:
Inclusion Criteria:

* About 80 single-rooted and premolar teeth with mature, fully formed apices and diagnosed with irreversible pulpitis will be selected.

Exclusion Criteria:

* Patients will be excluded if they were <12 years of age; pregnant; had an indication for antibiotic prophylaxis; uncontrolled hypertension or diabetes mellitus; chronic renal failure; hematologic diseases; HIV; osteoporosis treated with bisphosphonates; steroid therapy >5mg/day of prednisolone and prior to head and neck irradiation therapy. We will also exclude teeth with abnormal root canal anatomy, with more than 26mm in length and with advanced periodontal disease.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-02-27 (Actual)

PRIMARY OUTCOMES:
Evaluation of postoperative pain change during the first 48 hours after treatment | first 48 hours after treatment
  All patients will receive a paper with a visual analogue scale, to score their pain from 0 to 10. None of the patients will have analgesics prescribed immediately after the treatment. They will be advised to not take any medication at any point of the follow-up. If they need some advice or analgesic medication, they will be able to contact with the investigator.
  The investigator will reach the patients after 8, 24 and 48 h, in order to ask their pain intensity and to ask if they need to take any analgesic to stop the pain. In case of any patient mentioning an important pain, it will be advised to take Ibuprofen 600mg every 6 hours, until the pain disappears. If any patient is allergic to non-steroidal anti-inflammatories, they will be advised to take paracetamol 1g and not take more than 4g per day. All the controls will be recorded on each patient's chart.

CONTACTS AND LOCATIONS:
Overall Officials: Cláudia Rodrigues, PhD, Study Chair — Faculdade de Medicina Dentária da Universidade do Porto
Locations (1):
- Faculdade de Medicina Dentária da Universidade do Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No